CLINICAL TRIAL: NCT01699711
Title: Normalization of dyrk1A and APP Function as an Approach to Improve Cognitive Performance and Decelerate AD Progression in DS Subjects: Epigallocatechin Gallate as Therapeutic Tool
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Rafael de la Torre, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TESDAD
Record Dates: First submitted 2012-09-26; First posted 2012-10-04 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Down Syndrome (DS)
Keywords: APP function (amyloid precursor protein, cognitive stimulation, alzheimer disease. program
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease | interventions — epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Supplement: Epigallocatechin-3-gallate (EGCG) (Active Comparator): EGCG normally works as a dietary supplement. EGCG administration in Down syndrome patients will result in an improvement of their cognitive performance. A daily oral dose containing 9 mg/kg (range 6.9-12.7) of EGCG is given during twelve months.
  Interventions: Dietary Supplement: Epigallocatechin-3-gallate (EGCG)
- Placebo (Placebo Comparator): No active treatment is given.
  Interventions: Dietary Supplement: Epigallocatechin-3-gallate (EGCG)

INTERVENTIONS:
Dietary Supplement: Epigallocatechin-3-gallate (EGCG) — EGCG administration in Down syndrome patients will result in an improvement of their cognitive performance. A daily oral dose containing 9 mg/kg (range 6.9-12.7) of EGCG is given during twelve months.

SUMMARY:
Epigallocatechin-3-gallate (EGCG), the major catechin in green tea, is postulated to modulate dual specificity tyrosine-phosphorylation-regulated kinase 1A (DYRK1A) and amyloid beta precursor protein (APP) gene overexpression in the brains of Down syndrome mouse models. The clinical study is aimed at demonstrating that normalization of Dyrk1A and APP functions is a therapeutic approach to improve cognitive performance and decelerate AD (Alzheimer's disease) like progression.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed of DS neurological disease, aged between 14-29 years.
* Have given the consent to participate (official custody).

Exclusion Criteria:

* Subjects with neurological disease other than DS, relevant medical disease, co-morbid mental disorder or currently taking any treatment that could interfere with cognitive function or alter any key biomarkers and biochemical parameters analyzed.
* Having suffered from any major illness or undergoing major surgery in the last three months before the study.
* Regular ingestion of medication in the month preceding the study (exceptions for single doses of symptomatic medication administered up to the week preceding the trial).
* Current ingestion of vitamin supplements or catechins or AINE in the two weeks preceding the study.
* History of gastrointestinal, hepatic or renal problems or any other cause that may alter processes of absorption, distribution, metabolism, or excretion of the drug, or that might suggest gastrointestinal irritation to drug.
* Subjects following a vegetarian diet.
* Practice of physical exercise for more than 2 hours per day or energy consume/consumption of more than 3000 kcal per week.

Ages: 14 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Evaluation | From predose baseline to 19 months (end of treatment)
  a.Intelligence Quotient [Kaufman (K-BIT)], b.Attention [Spatial Span direct series (SSP), Choice Reaction Time (CRT) CANTAB battery]c. Psychomotor Speed [ (MOT) CANTAB battery] d.Episodic Memory [visuospatial: Paired Associates Learning (PAL) and visual: Pattern Recognition Memory (PRM) CANTAB battery; visuospatial learning Cued Recall Test (CRT) ] e.Executive Functions [working memory: SSP CANTAB battery; verbal semantic fluency; inhibition: Cats and Dogs; planning: Tower of London-Drexel (TOLDX) mental flexibility: Weigl Card Sorting Test ] f.Language:[ Expressive language: Boston naming test (BNT) ; Receptive language: Token Test (TT) g.Functional, quality of life and neuropsychiatric evaluation [Adaptative Behaviour Assessment System (ABAS-II): Dementia Questionnaire for People with Intellectual Disabilities (DMR): Neuropsychiatric Inventory (NPI); quality of life: Kidscreen; semi-structured interview to evaluate subjective effects concerning relevant changes.
Change in Amyloidosis Biomarkers | From predose baseline to 19 months (end of treatment)
  APP derived amyloid peptides in plasma (INNO-BIA)

SECONDARY OUTCOMES:
Treatment compliance | Predose baseline 3, 7, 13 months
Change in Biomarkers of lipid oxidation | Predose baseline: 3, 7, 13 months
  LDL (Low density lipoproteins), HDL (High density lipoprotein, cholesterol, triglycerides oxidized-LDL (Pentra Autoanalyzer, and ELISA Mercodia for LDLox
Change in DYRK1A activity biomarkers | Predose baseline 4 , 7 and 13 and 19 moths (end of treatment plus 6 months).
  Plasma homocysteine (Abbot AxyM), transthyretrin (ELISA) FOXO1 (DNA-binding ELISA nuclear extract from lymphocytes)
COMT val158met genetic polymorphism (catechol methyl transferase) (Taqman) | Predose baseline
Change in AST (SGOT -serum glutamic oxaloacetic transaminase-) and ALT (SGPT- Serum Glutamic Pyruvate Transaminase-) (Pentra Autoanalyzer, and ELISA Mercodia for LDLox) | Predose baseline 4 , 7 and 13 and 19 moths (end of treatment plus 6 months).
Change in Body Composition by electrical impedance (TANITA-MC-180) | Predose baseline 4 , 7 and 13 and 19 moths (end of treatment plus 6 months).
Changes in Neurophysiology | Predose baseline: 7, 13 months
  Parameters to be evaluated: (i) Motor threshold at Rest (MTR) for the Abductor Pollicis Brevis ( APB) muscle determination (ii) Basal single pulse response at rest for the APB at 110 of the MTR required, and (iii) Percentage of increase and decrease of the amplitude of the APB after double pulse, short and long pulse interval after transcranial magnetic stimulation (TMS).
Changes in Neuroimaging | Predose baseline: 7, 13 months
  Regional brain morphology and volume (FLAIR) sequence to assess possible white matter tissue macroscopic lesions), brain function in disease-specific neural systems: Intrinsic functional organization (i.e., functional connectivity) in the resting-state within the neural systems.

CONTACTS AND LOCATIONS:
Locations (1):
- IMIM (Institut Hospital del Mar d'Investigacions Mèdiques), Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] de la Torre R, de Sola S, Hernandez G, Farre M, Pujol J, Rodriguez J, Espadaler JM, Langohr K, Cuenca-Royo A, Principe A, Xicota L, Janel N, Catuara-Solarz S, Sanchez-Benavides G, Blehaut H, Duenas-Espin I, Del Hoyo L, Benejam B, Blanco-Hinojo L, Videla S, Fito M, Delabar JM, Dierssen M; TESDAD study group. Safety and efficacy of cognitive training plus epigallocatechin-3-gallate in young adults with Down's syndrome (TESDAD): a double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Neurol. 2016 Jul;15(8):801-810. doi: 10.1016/S1474-4422(16)30034-5. PMID 27302362